CLINICAL TRIAL: NCT07079358
Title: Improving Veteran Referral to Cardiac Rehabilitation: A Hybrid Effectiveness-Implementation Trial
Brief Title: Improving Veteran Referral to Cardiac Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 23-171
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Disease; Cardiac Rehabilitation
Keywords: Cardiac Rehabilitation; Hybrid Effectiveness-Implementation Trial
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A single-arm, pre-post intervention study comparing cardiac rehabilitation referral rates 6 months before and 6 months after implementing the Veterans Cardiac Rehabilitation Referral Program (VCR2P) at three VA medical centers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Veterans Cardiac Rehabilitation Referral Program (Experimental): All eligible Veterans hospitalized with cardiac rehabilitation-eligible conditions (acute myocardial infarction, coronary artery bypass grafting, percutaneous coronary intervention, cardiac valve surgery, or systolic heart failure) will receive the VCR2P intervention.
  Interventions: Behavioral: Veterans Cardiac Rehabilitation Referral Program

INTERVENTIONS:
Behavioral: Veterans Cardiac Rehabilitation Referral Program — 1. A CDS tool that identifies Veterans hospitalized with CR-eligible conditions and prompts physicians to refer them to CR.
  2. Educational materials that explain to Veterans the benefits and importance of participating in CR.
  3. Defined responsibilities for a facility-based CR referral coordinator who will support development and oversight of the referral process.

SUMMARY:
This study will test whether the Veterans Cardiac Rehabilitation Referral Program (VCR2P) improves cardiac rehabilitation participation by studying 816 Veterans across three VA medical centers in Nashville, Dallas, and Gainesville over 12 months. The trial compares referral rates from the 6 months before implementing the program to 6 months after, using a "before and after" design since randomization would be impractical. The study will measure whether the program increases the proportion of eligible Veterans who receive cardiac rehabilitation referrals and whether more Veterans actually attend rehabilitation sessions. Additionally, focus groups with physicians, nurses, and Veterans will identify what helps or hinders the program's success, providing essential insights for expanding this intervention to other VA facilities nationwide if it proves effective.

DETAILED DESCRIPTION:
This study seeks to evaluate the Veterans Cardiac Rehabilitation Referral Program (VCR2P) using a type 2 hybrid effectiveness-implementation design. The trial involves a single-arm, pre-post trial at three VA medical centers, enrolling a total of 816 Veterans who are eligible for cardiac rehabilitation (CR). The primary objective is to assess the program's impact on two key outcomes: CR referral rates and CR initiation rates. Secondary implementation outcomes will include measures such as reach, adoption, fidelity, maintenance, and cost, providing a comprehensive understanding of how the intervention performs in real-world VA settings. This evaluation will be guided by implementation science frameworks to ensure the program is scalable and sustainable. A summative evaluation will be conducted to inform broader implementation across the Veterans Health Administration. The goal is to determine not only whether VCR2P improves referral and participation in CR but also how it can be feasibly integrated into routine care to close quality gaps and enhance cardiovascular outcomes for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* All Veterans hospitalized with acute myocardial infarction, percutaneous coronary intervention, cardiac valve surgery, coronary artery bypass grafting, or systolic heart failure at the three participating VA medical centers (Nashville, Dallas, and Gainesville).

Exclusion Criteria:

* No exclusion criteria during the intervention period

  * however, post-hoc analysis will exclude Veterans with documented reasons preventing CR attendance including death during hospitalization or within 30 days of discharge, discharge to inpatient rehabilitation or skilled nursing facilities, significant cognitive impairment, high-risk ventricular arrhythmias, or explicit refusal of CR services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 816 (Estimated)
Dates: Start 2027-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac rehabilitation referral | From hospital admission to 30 days after discharge
  Proportion of eligible Veterans referred to cardiac rehabilitation.

SECONDARY OUTCOMES:
Cardiac rehabilitation initiation | Within 6 months of hospital discharge
  Proportion of eligible Veterans attending at least one cardiac rehabilitation session.

CONTACTS AND LOCATIONS:
Overall Officials: Justin M Bachmann, MD MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (3):
- United States (3):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No